CLINICAL TRIAL: NCT00004375
Title: Ultraviolet Light Therapy for Systemic Lupus Erythematosus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other)
Purpose: Treatment
Other Study IDs: NCRR-M01RR05096-0002; LSUMC-1765; LSUMC-910067
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: arthritis & connective tissue diseases; immunologic disorders and infectious disorders; rare disease; systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis; Connective Tissue Diseases; Immune System Diseases; Communicable Diseases; Rare Diseases

INTERVENTIONS:
Procedure: ultraviolet A-1 light treatment

SUMMARY:
OBJECTIVES:

I. Evaluate the mechanisms of ultraviolet A-1 light therapy in patients with systemic lupus erythematosus and normal controls.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Treatment with ultraviolet A-1 light is administered 5 days a week for 6 weeks, at the lowest dose or frequency required to maintain a response. The dose and frequency are progressively decreased over the next 9 weeks.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Patients ages 15 to 70 with symptomatic systemic lupus erythematosus meeting American Rheumatism Association criteria and normal controls

--Prior/Concurrent Therapy--

No requirement for tetracycline or other photosensitizing drugs

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 1991-09

CONTACTS AND LOCATIONS:
Overall Officials: Hugh McGrath, Jr., Study Chair — Louisiana State University Health Sciences Center in New Orleans
Locations (2):
- United States (2):
  - General Clinical Research Center and Charity Hospital (University of Louisiana), New Orleans, Louisiana
  - Alton Ochsner Medical Foundation Hospital, New Orleans, Louisiana

REFERENCES:
- [Background] McGrath H, Martinez-Osuna P, Lee FA. Ultraviolet-A1 (340-400 nm) irradiation therapy in systemic lupus erythematosus. Lupus. 1996 Aug;5(4):269-74. doi: 10.1177/096120339600500405. PMID 8869897